CLINICAL TRIAL: NCT03422835
Title: A Prospective Cohort Study of Robotic Transanal Total Mesentery Excision Versus Conventional Robotic Surgery for Rectal Cancer in Low Site
Brief Title: Robotic Assisted Transanal Total Mesorectal Excision Surgery for Rectal Cancer in Low Site
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, fan li, Prof., Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RATERAL-01
Record Dates: First submitted 2018-01-24; First posted 2018-02-06 (Actual); Last update posted 2018-02-06 (Actual); Status verified 2018-01

CONDITIONS: Rectal Neoplasms
Keywords: transanal surgery; robotic surgery; total mesorectal excision
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- R-TME (Active Comparator): Robotic total mesentery excision surgery for rectal cancer.
  Interventions: Procedure: R-TME
- R-TaTME (Experimental): Robotic transanal total mesentery excision surgery for rectal cancer.
  Interventions: Procedure: R-TaTME

INTERVENTIONS:
Procedure: R-TME — Conventional Robotic Total Mesentery Excision
  Arms: R-TME
Procedure: R-TaTME — Robotic Transanal Total Mesentery Excision
  Arms: R-TaTME

SUMMARY:
To investigates the feasibility, practicability, safety and subjective as well as functional outcome of Robotic transanal total mesentery excision for rectal cancer in low site.

DETAILED DESCRIPTION:
Transanal total mesorectal excision (TaTME) may offer a better way to achieve radical resection and functional protection for lower rectal cancer, which have been regarded as challenging situations in rectal cancer surgery. However, the narrow angle and limited space of the operation restrict the wide spread of this technique. Da Vinci robotic system has achieved good results in rectal cancer surgery. Robotics may help to overcome technical difficulties in TaTME. The purpose of this study was to explore the availability of Da Vinci robotic-assisted transanal total mesorectal excision(R-TaTME) This study investigates the feasibility, practicability, safety and subjective as well as functional outcome of Robotic transanal total mesentery excision for rectal cancer in low site.

ELIGIBILITY:
Inclusion Criteria:

* adenocarcinoma of the rectum by biopsy
* the lower edge of the tumor from the anal margin less than 8cm according to MRI or rigid endoscopy
* tumor diameter less than 4cm
* baseline clinical stage I-III: cT1-3 N0-2 M0 (AJCC v7)
* tolerable to surgery
* be able to understand and willing to participate in this trial with signature

Exclusion Criteria:

* history of malignant colorectal neoplasia
* recent diagnosis with other malignancies
* patients requiring emergency surgery such as obstruction，perforation and bleeding
* tumor involving adjacent organs, anal sphincter, or levator ani muscle muti-focal colorectal cancer
* preoperative poor anal function, anal stenosis, anal injury, or fecal incontinence history of inflammatory bowel disease or familial adenomatous polyposis
* participating in other clinical trails
* History of pelvic radiation
* BMI > 40
* Large uterine fibroids
* can not tolerate the surgery
* history of serious mental illness
* pregnancy or lactating women
* preoperative uncontrolled infection
* the researchers believe the patients should not enrolled in

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-02-15 (Estimated); Primary Completion 2020-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Positive rate of circumferential resection margin (CRM) of the specimens | 10 days after surgery
  Circumferential resection margin (CRM) is the distance between the deepest point of tumor in the primary cancer and the margin of resection in the retroperitoneum or mesentery by pathological examination. CRM 0-1mm is defined as positive, while >1mm is negative.

SECONDARY OUTCOMES:
The grade score of the specimens integrity | 10 days after surgery
  the quality of the specimens: grade 1 is bad gross specimen which means incomplete mesorectum and pelvic fascia, and muscle layer can be see >5mm; grade 3 is high quality gross specimen, which means the specimen is cylindrical, mesorectum and pelvic fascia are complete; grade 2 is between 1and 3.
The distance between lower tumor margin and the lower reaction margin | 10 days after surgery
  the oncological safety of the surgery by pathological examination. Reports should contain the distance between lower tumor margin and the lower reaction margin.
postoperative hospital stay | 3 years after surgery
  recovery information.
disease free survival rate | 3 years after surgery
  the oncological efficacy by 3-year follow-up according to the NCCN guideline. Participants should report every follow-up examinations which prove tumor recurrence and/or metastasis or not.
overall survival rate | 3 years after surgery
  the oncological efficacy by 3-year follow-up according to the NCCN guideline. Participants should report every follow-up examinations which prove tumor recurrence and/or metastasis or not.
the rate of postoperative complications | 30 days after surgery
  preoperative safety containing operation information, complication information.

OTHER OUTCOMES:
defecating functional outcomes | 3 years after surgery
  Wexner scale
sexual functional outcomes | 2 years after surgery
  We examine before operation, 3 months after, 6 months after, 12 months after, 24 months after operation, by questionnaires (International Index of Erectile Function (IIEF)
Quality of life outcomes evaluation | 2 years rafter surgery
  We examine before operation, 3 months after, 6 months after, 12 months after, 24 months after operation, by questionnaires (Short Form-36 (SF36).

CONTACTS AND LOCATIONS:
Overall Officials: fan li, MD., Principal Investigator — Daping Hospital, Third Military Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heald RJ, Husband EM, Ryall RD. The mesorectum in rectal cancer surgery--the clue to pelvic recurrence? Br J Surg. 1982 Oct;69(10):613-6. doi: 10.1002/bjs.1800691019. PMID 6751457
- [Background] Kim MJ, Park SC, Park JW, Chang HJ, Kim DY, Nam BH, Sohn DK, Oh JH. Robot-assisted Versus Laparoscopic Surgery for Rectal Cancer: A Phase II Open Label Prospective Randomized Controlled Trial. Ann Surg. 2018 Feb;267(2):243-251. doi: 10.1097/SLA.0000000000002321. PMID 28549014
- [Background] Kuo LJ, Ngu JC, Tong YS, Chen CC. Combined robotic transanal total mesorectal excision (R-taTME) and single-site plus one-port (R-SSPO) technique for ultra-low rectal surgery-initial experience with a new operation approach. Int J Colorectal Dis. 2017 Feb;32(2):249-254. doi: 10.1007/s00384-016-2686-3. Epub 2016 Oct 15. PMID 27744632
- [Background] Wang Y, Liu R, Zhang Z, Xue Q, Yan J, Yu J, Liu H, Zhao L, Mou T, Deng H, Li G. A safety study of transumbilical single incision versus conventional laparoscopic surgery for colorectal cancer: study protocol for a randomized controlled trial. Trials. 2015 Nov 30;16:539. doi: 10.1186/s13063-015-1067-5. PMID 26620555
- [Background] Odermatt M, Flashman K, Khan J, Parvaiz A. Laparoscopic-assisted abdominoperineal resection for low rectal cancer provides a shorter length of hospital stay while not affecting the recurrence or survival: a propensity score-matched analysis. Surg Today. 2016 Jul;46(7):798-806. doi: 10.1007/s00595-015-1244-x. Epub 2015 Sep 5. PMID 26342816
- [Background] Zhang H, Zhang YS, Jin XW, Li MZ, Fan JS, Yang ZH. Transanal single-port laparoscopic total mesorectal excision in the treatment of rectal cancer. Tech Coloproctol. 2013 Feb;17(1):117-23. doi: 10.1007/s10151-012-0882-x. Epub 2012 Aug 31. PMID 22936590
- [Background] de Lacy AM, Rattner DW, Adelsdorfer C, Tasende MM, Fernandez M, Delgado S, Sylla P, Martinez-Palli G. Transanal natural orifice transluminal endoscopic surgery (NOTES) rectal resection: "down-to-up" total mesorectal excision (TME)--short-term outcomes in the first 20 cases. Surg Endosc. 2013 Sep;27(9):3165-72. doi: 10.1007/s00464-013-2872-0. Epub 2013 Mar 22. PMID 23519489
- [Background] Fernandez-Hevia M, Delgado S, Castells A, Tasende M, Momblan D, Diaz del Gobbo G, DeLacy B, Balust J, Lacy AM. Transanal total mesorectal excision in rectal cancer: short-term outcomes in comparison with laparoscopic surgery. Ann Surg. 2015 Feb;261(2):221-7. doi: 10.1097/SLA.0000000000000865. PMID 25185463